CLINICAL TRIAL: NCT05803499
Title: Developing a Targeted Intervention for Sleep Disturbance in Spousal Bereavement
Brief Title: Rest to Overcome Loss and Reduce Risk
Acronym: RESTore Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Diana Chirinos-Downie, Assistant Professor of Preventive Medicine (Epidemiology), Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP0058437; STU00212514 (Other: Northwestern University Institutional Review Board); 5K01HL149987-02 (NIH)
Record Dates: First submitted 2023-02-21; First posted 2023-04-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Sleep Disturbance; Inflammation; Quality of Life; Bereavement; Spouses
Keywords: sleep disturbance; inflammation; quality of life; bereavement; spouses
MeSH Terms: conditions — Parasomnias; Inflammation

STUDY DESIGN:
Intervention Model Description: This pilot will test the targeted intervention for feasibility, acceptability, and preliminary effects. Participants will be randomized to either 1) the targeted intervention for bereavement and sleep disturbance based on Cognitive Behavior Therapy for Insomnia (CBT-I), and 2) an information-only control. Participants will complete self-report measures and an in-person visit at baseline and post-treatment, and a 6-month follow-up (psychosocial measures only).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will not be informed which arm they have been randomized into. Research assistants will also be blinded to randomization. Only the control and intervention session facilitators and Principal Investigator will be aware of participants' study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted Intervention for Sleep and Bereavement (Targeted CBT-I) (Experimental): This intervention consists of 6, 50-60-minute online individual sessions delivered via video conference. Content will include a CBT-I based program adapted to the specific needs of spousally bereaved individuals.
  Interventions: Behavioral: Targeted Cognitive Behavior Therapy for Insomnia
- Information-Only Control (Placebo Comparator): The information-only control consists of 1, 50-60-minute online individual session delivered via video conference. Content will provide basic psychoeducation about sleep and aging.
  Interventions: Other: Information-Only Control

INTERVENTIONS:
Behavioral: Targeted Cognitive Behavior Therapy for Insomnia — This intervention consists of six, 50-min. online individual sessions delivered via video conference. Content was developed by tailoring standard cognitive behavioral therapy for insomnia (CBT-I) to the specific needs of people who recently lost spouses/long-term partners, by using qualitative data gathered in focus groups. The intervention incorporates key concepts of CBT-I (sleep restriction; stimulus control) and positive emotion psychology (everyday mindfulness; gratitude and self-compassion). Individualized sleep plans (including weekly sleep windows) will be created for intervention participants, and each weekly session will involve a discussion about participants' progress in improving sleep disturbance. Support and recommended coping skills for loss and bereavement will also be provided.
  Arms: Targeted Intervention for Sleep and Bereavement (Targeted CBT-I)
Other: Information-Only Control — The control session (approx. 50-min. in length) will be delivered online in a one-to-one format (participant and facilitator) via videoconference. Educational brochures based on recommendations provided by the American Academy of Sleep Medicine focused on sleep and health and sleep hygiene education will be used. No specific or individualized recommendations will be given to control participants.
  Arms: Information-Only Control

SUMMARY:
The purpose of this study is to develop and optimize a targeted behavioral intervention for sleep disturbance among individuals who have recently lost a spouse/long-term cohabitating partner. In the first phase of this study, patient focus groups were conducted to gather information about the unique sleep challenges experienced by spousally bereaved individuals and the kinds of support they would like to receive from a program based on Cognitive Behavior Therapy for Insomnia (CBT-I). In the second phase of the study, a two-arm randomized controlled trial will be conducted to compare changes in sleep and inflammation among participants in the targeted CBT-I intervention to those in an information-only control. Participants will be asked to attend two in-person visits (at baseline and, approx. 8 weeks later, at post-treatment) to provide a blood sample and have vital signs and basic anthropometric measurements (height, weight, waist circumference) taken. After their baseline visit, participants will be randomized into either the targeted CBT-I intervention or the information-only control. The targeted CBT-I intervention will entail 6 online sessions (approx. 50 mins. each) delivered via videoconference by a trained facilitator, once per week over the course of approx. 6 weeks. The information-only control will entail 1 online session (approx. 50 mins.) delivered via videoconference by a trained facilitator. Sleep data (collected via both actigraphy watches and patient self-report sleep diaries) and data on mood, grief, and sleep habits will be collected from participants at three timepoints (baseline, post-treatment, and then again at a 6-month follow-up).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Has experienced the loss of a spouse/long-term cohabitating partner (i.e., partner who lived with participant for at least 1 year before passing) within the past 3 months
* Scores 5 or above on the Pittsburgh Sleep Quality Inventory (PSQI; administered by research staff during phone screening call)
* Must have access to an internet-enabled device (e.g., smartphone, computer, tablet) to take part in the online intervention

Exclusion Criteria:

* Under age 18
* Non-English speakers
* Those with a previously diagnosed sleep disorder (e.g., restless leg syndrome; note: individuals with obstructive sleep apnea (OSA) will be eligible as long as they use a continuous positive airway pressure (CPAP) machine at least 5 days a week for at least 5 hours per day)
* Those who have been taking prescribed sleep medication(s) for 6 months or more
* Those with autoimmune or inflammatory diseases (such as: acute or chronic immune system medical conditions, medications or other conditions that impact immune function (e.g., chronic fatigue syndrome [CFS], lupus, rheumatoid arthritis, Sjogren's disease, systemic lupus erythematosus [SLE], Hepatitis C, or any other immunosuppressive treatment requiring conditions, per investigator discretion).
* Those who regularly use illegal substances.
* Those who are on medications with major immunological consequences (e.g. steroids)
* Women who are pregnant or nursing
* Those who have been vaccinated in the past two weeks (note: these individuals may simply delay enrollment by two weeks if otherwise eligible)
* Those with significant visual or auditory impairment, medical or psychiatric condition that is unstable, requires immediate treatment or is judged to interfere with study protocol (e.g., substance abuse, psychotic disorder, cognitive disorder, current suicidal ideation)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | Approximately 18 months
  Feasibility of recruitment will be demonstrated by an enrollment benchmark of 2 participants per month.
Feasibility of recruitment | Approx. 18 months
  Feasibility of recruitment will also be measured by the proportion of eligible participants who are enrolled (consented) and randomized.
Adherence to the intervention | Approx. 6 months
  Adherence to the intervention will be measured by the number of sessions attended by participants.
Treatment-specific retention rates | Approx. 6 months
  Treatment-specific retention will be measured by the percentage of participants who complete the post-treatment assessment in each arm.
Acceptability | Approx. 6 months
  The acceptability of the intervention will be demonstrated by ≥ 85% completion of the study protocol across the sample.
Attrition | Approx. 6 months
  Attrition will be measured at each follow-up visit (post intervention and 6-month follow-up) and will be defined by the percentage of randomized participants who did not attend the follow-up visit. Causes of attrition will be measured by analyzing reasons for participant drop-out as documented over the course of the study.
Treatment-specific acceptability | Approx. 6 months
  Treatment-specific acceptability will be measured by preference ratings gathered during the post-treatment debriefing session for each arm.
Preliminary change in sleep disturbance | Approx. 6 months
  Using the previously validated Pittsburgh Sleep Quality Index (PSQI), change in sleep disturbance will be assessed from baseline to 1. post-intervention (6-8 weeks later), and a 2. six-month follow-up. Global scores on the PSQI range from 0 to 21, with a higher score indicating more severe sleep disturbance.

SECONDARY OUTCOMES:
Preliminary change in inflammation | Approx. 8 weeks
  Changes in inflammation will be measured via inflammatory marker values in participant blood samples (interleukin 6 [IL-6], interleukin 8 [IL-8], interleukin 10 [IL-10], tumor necrosis factor alpha [TNF-α]) and will be assessed from baseline to post-intervention (6-8 weeks later).
Preliminary change in quality of life | Approx. 6 months
  Using the previously validated Research and Development (RAND) Corporation 36-Item Short Form Health Survey (SF-36), change in self-reported quality of life (General Health Subscale) will be assessed from baseline to 1. post-intervention (6-8 weeks later), and a 2. six-month follow-up. The General Health Subscale of the SF-36 ranges from 0 to 100 with higher scores indicating more favorable quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the primary results of the trial after deidentification will be shared.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following publication of the primary results.
Access Criteria: Data will be available for individual participant data meta-analysis. Proposals may be submitted up to 36 months following publication of the primary results and should be directed to diana.chirinos@northwestern.edu.